CLINICAL TRIAL: NCT04417491
Title: Influence of Patient Expectations on Dry Needling Effects on Pain Outcomes in Mechanical Neck Pain
Brief Title: Patient Expectations and Dry Needling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Full Proffessor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URJC5006
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Neck Pain
Keywords: Neck Pain; Needling; Expectance
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (Experimental): The intervention group will receive real dry needling (fast in and fast out needling technique) in an active MTrP within upper trapezius muscle.
  Interventions: Device: Dry Needling
- Sham Needling (Sham Comparator): The placebo group will receive sham needling in an active MTrP within the upper trapezius muscle. A sham needle will be used as placebo. This needle has a blunt tip and retractable handle that created the illusion of a needle penetrating the skin.
  Interventions: Device: Sham Needling

INTERVENTIONS:
Device: Dry Needling — Real dry needling will be conducted according to the fast-in and fast-out principle. The intervention will be applied until a total of four local twitch responses will be elicited
  Arms: Dry Needling
Device: Sham Needling — Sham dry needling with be conducted with a sham needle device. This needle has a blunt tip and retractable handle that created the illusion of a needle penetrating the skin. When this needle touches the skin, a pricking sensation will be created. However, when pressure will be increased, the shaft of the needle disappears into the handle creating a sensation on the patient
  Arms: Sham Needling

SUMMARY:
Dry needling (DN) is a treatment technique used for treating musculoskeletal pain conditions. DN has shown to be effective on pain and function in patients with mechanical neck pain. Potential effects of DN can be related to several mechanisms, including physical, cognitive and emotional factors. This study will evaluate the role of the patient expectances related to the evolution (progress) of the condition, in this case, mechanical neck pain, in the effects of real or sham dry needling in sensitivity outcomes such as pain intensity or pressure pain sensitivity. Expectation of each patient in both groups will be considered positive, neutral or negative based on the outcomes of the Patient Shoulder Expectancies (PSOE) questionnaire which was adapted to the cervical spine.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific mechanical neck pain of at least 3 months of duration
* At least one active trigger point in the upper trapezius muscle which referred pain reproduces the neck pain symptoms

Exclusion Criteria:

* whiplash injury;
* previous cervical or thoracic surgery;
* cervical radiculopathy or myelopathy;
* diagnosis of fibromyalgia syndrome;
* having undergone physical therapy in the previous 6 months;
* fear to needles

Ages: 18 Months to 65 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-28 (Actual)

PRIMARY OUTCOMES:
Changes in Neck Pain Intensity between baseline and follow-up periods | Baseline, immediately after and 1 week after intervention
  The intensity of neck pain at rest and during active movement of the cervical spine in rotation will be assessed with a visual analogue scale (VAS).

SECONDARY OUTCOMES:
Changes in Pressure pain sensitivity between baseline and follow-up periods | Baseline, immediately after and 1 week after intervention
  Pressure pain thresholds (PPT) will be assessed at the upper trapezius muscle, spinous process of C7 and distant pain-free area of the lower extremity (heel)
Changes in patients self-perceived improvement between baseline and follow-up periods | Baseline and 1 week after intervention
  Patients self-perceived improvement will be assessed using a Global Rating of Change (GROC) consisting of a 15-point scale ranging from -7 (a very great deal worse) to +7 (a very great deal better).

CONTACTS AND LOCATIONS:
Locations (1):
- César Fernández-de-las-Peñas, Alcorcón, Rest of the World, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gallego-Sendarrubias GM, Voogt L, Arias-Buria JL, Bialosky J, Fernandez-de-Las-Penas C. Can Patient Expectations Modulate the Short-Term Effects of Dry Needling on Sensitivity Outcomes in Patients with Mechanical Neck Pain? A Randomized Clinical Trial. Pain Med. 2022 May 4;23(5):965-976. doi: 10.1093/pm/pnab134. PMID 33830234